CLINICAL TRIAL: NCT03022461
Title: HeartMate 3 CE Mark Study Long Term Follow-up Clinical Investigation Plan
Brief Title: HeartMate 3 CE Mark Study Long Term Follow-up
Acronym: HM3 CE LTFU
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: HeartMate 3 CE Mark Study LTFU
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure
Keywords: Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Disease; Cardiovascular Disease; Heart-assist Devices; Thoratec Corporation
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ongoing HM3 CE Mark study patients: The study will include the ongoing HM3 CE Mark study patients that have consented to continue the long term follow-up data collection.
  Interventions: Other: Long term follow-up

INTERVENTIONS:
Other: Long term follow-up

SUMMARY:
The purpose of this clinical investigation is to report the long term survival and incidence of adverse events in the patients who were implanted with HM3 in the CE Mark Study and continue to be ongoing with the HeartMate 3 LVAS after the CE Mark Study 2 year follow-up.

The study will be a single arm, prospective, multi-center, non-blinded and non-randomized study, intended to report on the long term use of the HeartMate 3 LVAS in those patients that completed the 2-year follow-up in the HeartMate 3 CE Mark study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative has signed Informed Consent Form (ICF).
2. Patient was enrolled in the HeartMate 3 CE Mark Study and continues to be supported with the HeartMate 3 LVAS after the 2 year CE Mark study follow-up.

Exclusion Criteria:

1. Patient does not consent to the continued data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced refractory left ventricular heart failure who were implanted with HeartMate 3 in the CE Mark Study and continue to be ongoing with the HeartMate 3 LVAS after the CE Mark Study 2 year follow-up will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gazzola, B. Sc., Study Director — Abbott
Locations (8):
- The Alfred Hospital, Melbourne, Victoria, Australia
- AKH Medical University of Vienna, Vienna, Austria
- Toronto General Hospital, Toronto, Ontario, Canada
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia
- Germany (3):
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitats-Herzzentrum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
- National Research Center for Cardiac Surgery, Astana, Kazakhstan

RESULTS

PARTICIPANT FLOW:
Groups:
- Ongoing HM3 CE Mark Study Patients: Patients who were ongoing after two years follow-up in the HeartMate 3 CE Mark study (NCT02170363) and consented to participate in long-term follow-up data collection.
Period: Overall Study
Arm/Group | Ongoing HM3 CE Mark Study Patients
Started | 25
Completed | 22
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 2
  Austria | 2
  Czechia | 7
  Kazakhstan | 4
  Australia | 1
  Germany | 9
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.0 (0.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (4.7)
Ischemic Etiology [Count of Participants; unit: Participants] | 11
Indication for Left Ventricular Assist Device (LVAD) implant [Count of Participants; unit: Participants]
  Bridge to cardiac transplantation (BTT) | 14
  Permanent destination therapy (DT) | 11
INTERMACS Profile [Count of Participants; unit: Participants] — INTERMACS profiles are scaled depending on the patients condition from 7 (clinically stable with a reasonable level of comfortable activity) to 1 (critical cardiogenic shock)
  Participants
    Profile 1 | 0
    Profile 2 | 1
    Profile 3 | 9
    Profile 4 | 14
    Profile 5 | 1
    Profile 6 | 0
    Profile 7 | 0
Cardiac Index [Mean (Standard Deviation); unit: l/min/m^2] — Cardiac index (CI) is a haemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA), thus relating heart performance to the size of the individual.
  l/min/m^2 | 1.7 (0.34)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percentage] — The ejection fraction (EF) is the volumetric fraction (or portion of the total) of fluid (usually blood) ejected from a chamber (usually the heart) with each contraction (or heartbeat). The left ventricular ejection fraction (LVEF), is calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume). LVEF is an indicator of the effectiveness of pumping into the systemic circulation.
  percentage | 19.4 (3.7)
Central Venous Pressure (CVP) [Mean (Standard Deviation); unit: mmHg] | 9.3 (5.01)
Arterial Blood Pressure [Mean (Standard Deviation); unit: mmHg] — The systolic pressure is the pressure during the heart contraction phase (systole) The mean arterial pressure is an average blood pressure in an individual during a single cardiac cycle The diastolic pressure is the pressure during the heart relaxation phase (diastole)
  mmHg
    Systolic pressure | 105.3 (11.7)
    Mean pressure | 77.5 (8.6)
    Diastolic pressure | 23.1 (9.5)
Pulmonary Artery Pressure [Mean (Standard Deviation); unit: mmHg] — The systolic pressure is the pressure during the heart contraction phase (systole) The mean arterial pressure is an average blood pressure in an individual during a single cardiac cycle The diastolic pressure is the pressure during the heart relaxation phase (diastole)
  mmHg
    Systolic | 51.8 (20.8)
    Mean | 33.7 (13.3)
    Diastolic | 23.1 (9.5)
Pulmonary Capillary Pressure [Mean (Standard Deviation); unit: mmHg] | 22.2 (10.1)
White Blood Cell count [Mean (Standard Deviation); unit: 10^3 cells/ml] | 7.2 (1.9)
Plasma-free Hemoglobin [Mean (Standard Deviation); unit: mg/dl] | 13.8 (16.3)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — The INR is the ratio of a patient's prothrombin time to a normal (control) sample, raised to the power of the ISI (International Sensitivity Index) value for the analytical system being used
  ratio | 1.36 (0.5)
Prothrombin time [Mean (Standard Deviation); unit: s] | 15.7 (4.6)
Partial thromboplastin time [Mean (Standard Deviation); unit: s] | 38.9 (5.8)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/l] | 4.1 (1.4)
Lactic Dehydrogenase (LDH) [Mean (Standard Deviation); unit: U/l] | 4.0 (1.0)
Medications [Count of Participants; unit: Participants]
  ACE Inhibitor | 12
  Angiotensin II antagonist | 5
  Beta-blocker | 17
  Anticoagulant/antiplatelet drug | 23
  Antiarrhythmic drug | 11
  Inotropes type 1 | 7
  Inotropes type 2 | 5
Pre-operative Risk Factors [Count of Participants; unit: Participants]
  Hypertension | 17
  Diabetes | 6
  Prior sternotomy | 6
  Severe Chronic Obstructive Pulmonary Disease (COPD) | 1
  Transient Ischemic Attack (TIA) | 3
  Stroke | 1
  Renal Dysfunction | 12
  Arrhythmia | 19
  Pacemaker/defibrillator | 19
  Valve disease | 21
  Peripheral vascular disease | 2
  Left ventricular aneurism | 3

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Subject outcomes and survival over time
Time Frame: At 5 years post HM3 CE Mark study implant
Measure: Number (95% Confidence Interval); unit: percentage of patients who survived
Groups:
- Ongoing HM3 CE Mark Study Patients: Ongoing HM3 CE Mark study (NCT02170363) patients that have consented to continue the long term follow-up data collection.
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
percentage of patients who survived | 61 [44 to 74]

2. Secondary Outcome: EuroQoL 5D-5L (EQ-5D-5L) VAS Score
Description: Quality of Life over time as measured by EuroQoL 5D-5L (EQ-5D-5L) VAS Score. The Visual Analog Scale (VAS) records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher quality of life
Time Frame: At 5 years post HM3 CE Mark study implant
Population: The population analyzed is composed by patients for whom the EQ-5D-5L questionnaire was available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 20
score on a scale | 69.3 (19.3)

3. Secondary Outcome: Six Minute Walk Test (6MWT)
Description: Functional status over time as measured by the Six Minute Walk Test (6MWT). The 6MWT is done to establish the amount of meters a subject can walk in 6 minutes
Time Frame: At 5 years post HM3 CE Mark study implant
Population: The population analyzed is composed by patients for whom the 6MWT was available
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 22
meters | 294.4 (155.8)

4. Secondary Outcome: New York Heart Association (NYHA)
Description: Functional status over time as measured by New York Heart Association (NYHA). Patients are graded from 4 to 1 in order or symptoms:
  I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  IIIA Marked limitation of physical activity. No dyspnea at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IIIB Marked limitation of physical activity. Recent dyspnea at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: At 5 years post HM3 CE Mark study implant
Population: The population analyzed is composed by patients for whom the NYHA class was available
Measure: Count of Participants; unit: Participants
Groups:
- Ongoing HM3 CE Mark Study Patients: Ongoing HM3 CE Mark study patients that have consented to continue the long term follow-up data collection.
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 21
Participants
  NYHA Class I | 9
  NYHA Class II | 10
  NYHA Class IIIA | 2
  NYHA Class IIIB | 0
  NYHA Class IV | 0

5. Secondary Outcome: Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: Between 2 and 5 years post HM3 CE Mark study implant
Population: Ongoing HM3 CE Mark study patients that have consented to continue the long term follow-up data collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
Participants
  Bleeding | 3
  Infection | 9
  Stroke, Ischemic | 2
  Stroke, Hemorrhagic | 3
  Pump Thrombosis | 0
  Hemolysis | 0
  Right Heart Failure | 1

6. Secondary Outcome: Device Malfunctions
Description: Number of Participants with device malfunctions
Time Frame: Between 2 and 5 years post HM3 CE Mark study implant
Measure: Number; unit: participants
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
participants | 0

7. Secondary Outcome: Reoperations
Description: Number of reoperations
Time Frame: Between 2 and 5 years post HM3 CE Mark study implant
Measure: Number; unit: events
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
events
  Major bleeding | 1
  Major infection | 6
  Neurologic dysfunction | 4
  Other Reoperation | 11

8. Secondary Outcome: Rehospitalizations
Description: Number of rehospitalizations
Time Frame: Between 2 and 5 years post HM3 CE Mark study implant
Measure: Number; unit: events
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
events
  Cardiac Arrhythmia | 1
  Infection | 19
  Bleeding | 2
  Neurological Event | 2
  Renal Dysfunction | 1
  Respiratory Insufficiency | 0
  Right Heart Failure | 1
  Other Adverse Event | 13

9. Secondary Outcome: Percentage of Participants Who Survived Without Experiencing a Debilitating Stroke (MRS>3)
Description: Modified Rankin Score >3 is considered debilitating. As in 3 cases the MRS evaluation was not available, a sensitivity analysis for the worst and best case scenario was performed.
  The MRS scale is as following:
  0: No observed neurological symptoms; 1: No significant neurological disability despite symptoms; able to carry out all usual duties and activities; 2: Slight neurological disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3: Moderate neurological disability; requiring some help, but able to walk without assistance; 4: Moderate severe neurological disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5: Severe neurological disability; bedridden, incontinent and requiring constant nursing care and attention as a result of a neurological deficit; 6: Dead
Time Frame: As it may occur up to 5 years post HM3 CE Mark study implant or to outcome, whichever occurs first
Population: In 3 cases the MRS evaluation was not available, a sensitivity analysis for the worst and best case scenario was performed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ongoing HM3 CE Mark Study Patients
Number analyzed (Participants) | 25
percentage of participants
  Assuming three patients with missing MRS had debilitating stroke | 55.1 [39.1 to 68.5]
  Assuming three patients with missing MRS had non-debilitating stroke | 61.0 [44.6 to 73.9]

ADVERSE EVENTS:
Time Frame: Events were collected as of 2 to 5 Years follow-up post implant
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device under investigation.
Arm/Group | Ongoing HM3 CE Mark Study Patients
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 13/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ongoing HM3 CE Mark Study Patients (N=25)
Pump Thrombosis (Product Issues) | 0
Bleeding (Vascular disorders) | 3
Hemolysis (Blood and lymphatic system disorders) | 0
Infection (Infections and infestations) | 9
Right Heart Failure (Cardiac disorders) | 1
Stroke, Hemorrhagic (Nervous system disorders) | 3
Stroke, Ischemic (Nervous system disorders) | 2
Cardiac Arrhythmia (Cardiac disorders) | 1
Renal Dysfunction (Renal and urinary disorders) | 1
Outflow Graft Thrombosis (Product Issues) | 2
Other Neurological event (Nervous system disorders) | 1
Pump Malfunction (Product Issues) | 0
Psychiatric Episode (Nervous system disorders) | 0
Hepatic Dysfunction (Hepatobiliary disorders) | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0
Hypertension (Vascular disorders) | 0
Pericardial Fluid Collection (Blood and lymphatic system disorders) | 0
Other Adverse Event (Cardiac disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT03022461/Prot_SAP_000.pdf